CLINICAL TRIAL: NCT05322811
Title: Emotional State Among Patients With Neurological Disorders
Status: Completed | Type: Observational
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Evgenia Trevlaki, Clinical Professor, International Hellenic University
Other Study IDs: InternationalHellenicU
Record Dates: First submitted 2022-02-03; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Emotional Stress; Emotional Depression; Anxiety; Neurologic Disorder
Keywords: stress; anxiety; depression; neurologic disorders
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adults patients with neurological disorder

SUMMARY:
The purpose of the study was to examine the emotional state of the patients with neurological disorders. The evaluation was conducted with DASS-21 scale over 40 patients.

DETAILED DESCRIPTION:
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.The DASS-21 should not be used to replace a face to face clinical interview.

ELIGIBILITY:
Inclusion Criteria:

* patients with neurological disorders

Exclusion Criteria:

* not given concent
* Incomplete questionaire answers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with neurological disorders
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Emotional state score of the patients | through study completion, an average of 1 year
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Scores on the DASS-21 will need to be multiplied by 2 to calculate the final score. Minimum score 0, maximum score 116+. The high score means a worse outcome.

SECONDARY OUTCOMES:
Stress frequency at the participants | through study completion, an average of 1 year
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Minimum score for stress is 0, maximum score 34+. The high score means a worse outcome.
Depression frequency at the participants | through study completion, an average of 1 year
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Minimum score for stress is 0, maximum score 28+. The high score means a worse outcome.
Anxiety frequency at the participants | through study completion, an average of 1 year
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Minimum score for stress is 0, maximum score 20+. The high score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra-Hristara Papadopoulou, Study Chair — PhD Professor of Physiotherapy at IHU, Head of the Postgraduate Programme, Pediatric Physiotherapy
Locations (1):
- Physical therapy clinic Trevlakis Emmanouil, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05322811/Prot_000.pdf